CLINICAL TRIAL: NCT03509116
Title: Understanding the Experience of the Dietetic Consultation and the Perceptions of Its Value From the Perspective of Nutritionally Vulnerable Older Patients, Dietitians and Other Key Stakeholders: an Illuminative Evaluation
Brief Title: The Dietetic Consultation: an Illuminative Evaluation
Status: Completed | Type: Observational
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: 184290
Record Dates: First submitted 2018-04-16; First posted 2018-04-26 (Actual); Results first posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-12

CONDITIONS: Malnutrition
Keywords: patient experience; disease-related malnutrition; nutritional care; dietetic consultation; older adults; oral nutritional support
MeSH Terms: conditions — Malnutrition | interventions — Watchful Waiting; Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patient group 1: Consultation observation, documentary analysis
  Interventions: Other: Observations, documents
- Patient group 2: Qualitative interview, key stakeholders, documentary analysis
  Interventions: Other: Interviews, key stakeholders, documents
- Dietitians: Consulting Dietitians
  Interventions: Other: Observations, documents; Other: Interviews, key stakeholders, documents
- Key Stakeholders: Patient-Nominated Key Stakeholders (Relatives/Carers)
  Interventions: Other: Interviews, key stakeholders, documents

INTERVENTIONS:
Other: Observations, documents — Consultation observations, documentary analysis
  Groups: Dietitians; Patient group 1
Other: Interviews, key stakeholders, documents — Qualitative interviews, key stakeholders, documentary analysis
  Groups: Dietitians; Key Stakeholders; Patient group 2

SUMMARY:
This study aims to understand the experience of the dietetic consultation from the perspective of nutritionally vulnerable older patients receiving oral nutrition support and dietitians, as well as other key stakeholders involved in the process of such a consultation.

Malnutrition is prevalent and increases the risk of health complications and socioeconomic burden. Patients with malnutrition are often older patients with complex needs and therefore may require specialist knowledge and skills to provide nutritional support. Dietitians are uniquely skilled to assess the multiple factors that underpin diet and to tailor nutritional support, which could help improve outcomes. Although the causes of malnutrition are complicated, its treatment typically involves oral nutritional supplements, dietary advice or food-based interventions, either separately or in combination.

Effectiveness of the various oral nutritional support interventions has been studied, with the findings on food-based interventions suggesting more research is needed and the widespread research on ONS suggesting contradictory results and interpretations. Despite this, the factors responsible for these inconsistencies have not been identified. There are no studies so far that have examined the patient experience of the consultation with the dietitian in the context of nutritional support. Although the patient experience of consultations is increasingly being recognised as an important part of investigating their effectiveness in healthcare, to date, there are a number of limitations in this literature, leaving the role of the patient experience in dietetic consultations for the management of malnutrition, poorly understood. It's probable that this is one contributing factor to the variation observed in the literature.

A review of the literature indicates a need for exploration of the patient experience and its possible impact on the success or failure of the dietetic encounter. This study aims to address some of the knowledge gaps. The use of qualitative interviews will allow an in-depth understanding of the experience of the dietetic consultation for the provision of nutrition support and will utilise an overall illuminative evaluation approach to broaden that understanding by considering data from various sources. Participants will include older patients who are considered nutritionally vulnerable, their consulting dietitians and patient-nominated key stakeholders. Four clinical settings within the Trust where dietitians would often see patients for nutritional support will be included.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Adults (aged > 60 years)
* National Health Service (NHS) number
* Capable of giving informed consent
* Able to communicate well in English
* Nutritionally vulnerable according to the Nutrition Screening Tool in use at the NHS Trust prompting referral to a dietitian
* Likely to receive a form of oral nutrition support in the management of malnutrition
* A variety of the patient characteristics detailed earlier will be included where possible
* Consents to having their qualitative interview audio-recorded (Group 2)

Dietitians:

* Consulting dietitian providing the nutritional advice to patient above
* Employee of the NHS Trust and member of the Nutrition & Dietetic team
* Minimum of three different dietitians across the healthcare settings to be included
* Consents to having their qualitative interview audio-recorded

Key Stakeholders:

Up to 2 optional patient-nominated key stakeholders who are involved in the dietetic consultation and success of the dietetic intervention e.g. other HCP, family member, carer or friend. Their criteria for inclusion will include:

* Nominated by the patient (from Group 2) participating in the study
* Involved in some aspect of the implementation of goals agreed between the patient and dietitian during the consultation i.e. the nutritional intervention
* Available for separate interview at a mutually agreed location
* Capable of giving informed consent
* Able to communicate well in English
* Consents to having their qualitative interview audio-recorded

Exclusion Criteria:

Patients:

* Participated or due to participate in another aspect of the study i.e. a patient will not be recruited to participate in consultation observations if they have already been or due to be recruited to take part in the qualitative interviews and vice versa.
* Outside of stated age range for inclusion
* Incapable of giving informed consent
* No National Health Service (NHS) number
* Unable to communicate well in English
* Not considered nutritionally vulnerable according to Nutrition Screening Tool
* Not referred to a dietitian for nutrition support
* Patients receiving artificial nutrition support
* Does not wish to have their qualitative interview audio-recorded (Group 2)

Participants with visual or hearing impairment or other physical disabilities will NOT be excluded from the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients:
  Older patients malnourished or at risk of malnutrition requiring oral nutritional support from a dietitian in a range of clinical settings.
  Dietitians:
  Consulting registered dietitian providing the nutritional advice to patient above
  Key Stakeholders:
  Up to 2 optional patient-nominated key stakeholders who are involved in the dietetic consultation and success of the dietetic intervention e.g. other HCP, carer or family member.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2022-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alastair Duncan, PhD, Study Chair — King's College London
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Please note that 45 participants were enrolled but only 39 took part in research activities. 4 dietitians gave consent but did not complete the study activities due to changes in their clinical speciality, change in employment, maternity leave and lack of eligible patients within the study time frame. Also, 2 patients gave consent but didn't complete the study activities, 1 patient died before this was possible and 1 withdrew their consent to participate so no research activities were commenced.
Groups:
- Key Stakeholders: Patient-nominated Key Stakeholders
Period: Overall Study
Arm/Group | Patient Group 1 | Patient Group 2 | Dietitians | Key Stakeholders
Started | 10 | 11 | 13 | 5
Completed | 10 | 11 | 13 | 5
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Key Stakeholders: Key stakeholders (relatives/carers of the patient.
- Total: Total of all reporting groups
Arm/Group | Patient Group 1 | Patient Group 2 | Dietitians | Key Stakeholders | Total
Number analyzed (Participants) | 10 | 11 | 13 | 5 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 13 | 2 | 15
  >=65 years | 10 | 11 | 0 | 3 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 7 | 11 | 5 | 26
  Male | 7 | 4 | 2 | 0 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 3 | 0 | 0 | 3
  White | 10 | 7 | 0 | 0 | 17
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 13 | 5 | 18
Region of Enrollment [Number; unit: participants]
  United Kingdom | 10 | 11 | 13 | 5 | 39
Clinical setting [Count of Participants; unit: Participants]
  Hospital | 6 | 3 | 6 | 1 | 16
  Outpatient clinic | 2 | 5 | 3 | 3 | 13
  Community | 2 | 3 | 4 | 1 | 10

OUTCOME MEASURES:

1. Primary Outcome: Experience of the Dietetic Consultation (Number of Participants With Dietetic Consultation Experience That Relate to Each Theme)
Description: Themes and sub-themes related to the patient experience, dietitian experience and key stakeholder experience of the consultation. These were derived from qualitative thematic analysis of triangulated data from interviews, consultation observations and consultation documents derived from ALL study participants (n=39). Final themes included: 1. Building a therapeutic alliance 2. Navigating changes beyond the consultation 3. Dynamics of expectations, power and satisfaction 4. Influences and realities of professional practice. Please note that ALL study participants (n=39) from all 4 groups (Patient Group 1, Patient Group 2, Dietitians, and Key Stakeholders) contributed to all 4 final constructed themes noted above as all data were qualitatively triangulated. These 4 themes represent how the dietetic consultation was experienced from multiple perspectives, in different contexts and highlighted key areas of the dietetic encounter that mattered to participants.
Time Frame: Through study completion, an average of 2 months
Measure: Count of Participants; unit: Participants
Groups:
- Patient Group 1: Number of participants for whom data were gathered from dietetic consultation observations and documentary analysis.
  Observations, documents: Consultation observations, documentary analysis
- Patient Group 2: Number of participants for whom data were gathered from qualitative interview, key stakeholders, and documentary analysis.
  Interviews, key stakeholders, documents: Qualitative interviews, key stakeholders, documentary analysis
- Dietitians: Number of participants who were consulting dietitians and for whom data were gathered from consultation observations and/or interviews and consultation documents.
- Key Stakeholders: Number of participants who were Patient-nominated Key Stakeholders and for whom data were gathered from consultation observations or interviews and consultation documents.
Arm/Group | Patient Group 1 | Patient Group 2 | Dietitians | Key Stakeholders
Number analyzed (Participants) | 10 | 11 | 13 | 5
Participants
  1. Building a therapeutic alliance | 10 | 11 | 13 | 5
  2. Navigating changes beyond the consultation | 10 | 11 | 13 | 5
  3. Dynamics of expectations, power and satisfaction | 10 | 11 | 13 | 5
  4. Influences and realities of professional practice | 10 | 11 | 13 | 5

2. Other Pre Specified Outcome: Dietitian AfC Banding
Description: The NHS AfC Banding for consulting dietitians included. NHS Band 5 = entry level dietitian, NHS Band 6 = more experienced and specialised dietitian, NHS Band 7 = more advanced level dietitian. Data were collected on the NHS Banding (determined by their employer) for each dietitian included to understand how their experiences differed by seniority. Data collected for dietitians only.
Time Frame: At enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | Dietitians
Number analyzed (Participants) | 13
Participants
  Band 5 | 3
  Band 6 | 6
  Band 7 | 4

3. Other Pre Specified Outcome: Dietitian Speciality
Description: Clinical speciality of consulting dietitians included. Data collected for dietitians only.
Time Frame: At enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Dietitians
Number analyzed (Participants) | 13
Participants
  Stroke / Elderly Care | 3
  Community | 4
  Oncology | 2
  General | 2
  Gastro | 0
  Renal | 2
  HIV | 0

4. Other Pre Specified Outcome: Type of Intervention
Description: Type of nutritional support intervention the patient received during dietetic consultation. Data collected for patients only.
Time Frame: At enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Group 1 | Patient Group 2
Number analyzed (Participants) | 10 | 11
Participants
  ONS only (Oral nutritional supplements only) | 0 | 2
  FB only (Food-based intervention only) | 0 | 0
  COMB intervention (ONS + FB) | 10 | 9

5. Other Pre Specified Outcome: Consultation Type
Description: New (i.e. new episode of dietetic care) or review/follow-up (had previous consultation in current episode of care) re the dietetic consultation. Data collected for patients only.
Time Frame: At enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Group 1 | Patient Group 2
Number analyzed (Participants) | 10 | 11
Participants
  New | 2 | 2
  Review/Follow-up | 8 | 9

6. Other Pre Specified Outcome: Family Support
Description: Whether the patient had family support or not at the time of study enrollment. Data collected for patients only.
Time Frame: At enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Group 1 | Patient Group 2
Number analyzed (Participants) | 10 | 11
Participants
  Yes | 7 | 9
  No | 3 | 2

7. Other Pre Specified Outcome: Relationship to Patient
Description: Relationship of key stakeholder to patient. Data collected for key stakeholders only.
Time Frame: At enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | Key Stakeholders
Number analyzed (Participants) | 5
Participants
  Spouse | 3
  Other relative | 2

ADVERSE EVENTS:
Time Frame: From participant recruitment date until the final date when their research activities were completed - on average < 3 months.
Description: Please note these data were not routinely collected unless the patient died after providing consent but before their research activity (consultation observation or qualitative interview) was completed.
Groups:
- Key Stakeholders: Patient-nonimated key stakeholders
Arm/Group | Patient Group 1 | Patient Group 2 | Dietitians | Key Stakeholders
All-Cause Mortality (participants affected / at risk) | 0/10 | 1/11 | 0/13 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11 | 0/13 | 0/5
Other Adverse Events (participants affected / at risk) | 0/10 | 0/11 | 0/13 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2020-01-21): https://cdn.clinicaltrials.gov/large-docs/16/NCT03509116/Prot_000.pdf